CLINICAL TRIAL: NCT04063748
Title: Leuven Interactive Scheme for hearingTraining Evaluation, and Audiological Rehabilitation
Acronym: LUISTER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Astrid Van Wieringen, PhD, Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S59845
Record Dates: First submitted 2019-08-10; First posted 2019-08-21 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Hearing Disability
Keywords: auditory rehabilitation

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either the test or the placebo group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant does not know whether (s)he receives treatment or placebo. The investigator and the outcomes assessor are blind to this information too. The care provide (speech therapist) would know after communication with the participant.
  In case of the HA-study, participants either receive an intervention or do not receive an intervention. Therefore, they cannot be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): Participants are asked to train (at least) 5 times a week during 15 - 20 mins. The first 4 sessions are training sessions, the fifth session is an in-training test session (DTT and phoneme discrimination).
  Interventions: Behavioral: Audiological rehabilitation
- Placebo (Other): CI-users: Participants are asked to train (at least) 5 times a week during 15 - 20 mins. The first 4 sessions are training sessions, and the fifth session is an in-training test session (DTT and phoneme discrimination).
  Interventions: Behavioral: Placebo Rehabilitation
- Passive Control (Placebo Comparator): HA users: Participants do not receive an intervention.
  Interventions: Behavioral: Passive Control

INTERVENTIONS:
Behavioral: Audiological rehabilitation — Experimental: tablet-based take-home auditory-cognitive training, which consists of phoneme tasks, words in quiet and in different types of noise
  Other Names: LUISTER
  Arms: Experimental
Behavioral: Placebo Rehabilitation — CI-users: Placebo, tablet-based take-home psychophysical tasks, reading (non auditory)
  Arms: Placebo
Behavioral: Passive Control — No intervention in the passive control group for HA-users.
  Arms: Passive Control

SUMMARY:
It is believed that persons with hearing impairment benefit from auditory rehabilitation (AR), i.e. regular assessment and training of their listening skills. However, the efficacy of auditory rehabilitation has not been investigated before. In Leuven (Belgium) an e-health app has been developed that enables performance assessment, listening skills training, and counselling for persons with hearing impairment. Currently, an RCT is prepared to evaluate the different modules in persons with hearing impairment. The experimental group will receive auditory rehabilitation training modules, and a control group will either receive training tasks that are NOT believed to transfer to improved listening skills or will not receive any training (passive control).

1. Do participants improve on the trained tasks in the LUISTER AR scheme and does this improvement transfer to an improvement in speech perception in noise (primary outcome), executive functioning and/or quality of life (secondary outcomes)?
2. Does training with the LUISTER AR scheme provide more benefit on primary and secondary outcomes than a placebo program (active control group) or no training (passive control group)?
3. Can improvement in speech in noise perception, obtained with the LUISTER AR scheme, be consolidated until 6 months after training has stopped?
4. Are certain user-specific or training-specific aspects correlated to improvement on task-specific learning as well as near- and far transfer

DETAILED DESCRIPTION:
Goals of the study:

To determine an optimal, personalized AR scheme (considering age, degree of HI) and possible interacting factors (e.g., training time, type of errors)

To investigate transfer of auditory and auditory-cognitive training to listening skills in everyday life

To develop evidence-based guidelines for clinical AR

A study to assess the efficacy in CI users will start with baseline assessment (speech in noise understanding, LIST sentences and cognitive tests (executive functioning, important for listening skills). This will be followed by 8 weeks of training, an intermediate assessment moment, again 8 weeks of training, and a final evaluation moment. After 6 months follow-up evaluation to investigate retention. This study is comprised of an active training group and an active control group.

A study to assess the efficacy in HA users will start with baseline assessment (speech in noise understanding, LIST sentences and cognitive tests (executive functioning, important for listening skills). This will be followed by 6 weeks of training, an intermediate (online) assessment moment, again 6 weeks of training, and a final evaluation moment.

ELIGIBILITY:
Inclusion Criteria:

* hearing impaired
* sufficient knowledge of the Dutch language

Exclusion Criteria:

* cognitively impaired

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Speech in noise intelligibility | Change at 16 wks compared to baseline
  LIST sentences presented in speech-weighted noise. Participants are required to repeat sentences in noise. The Leuven Intelligibility Sentences Test (LIST, (van Wieringen & Wouters, 2008)) was specifically designed for speech perception in noise assessment in CI users. The test has a high test-retest reliability and a steep slope making it very sensitive to small improvements in performance.
  An improvement of 2dB results in a clinically relevant improvement in speech. discrimination in noise. Therefore, the primary endpoint to validate the LUISTER AR scheme will be an improvement of 2dB on speech discrimination in noise.

SECONDARY OUTCOMES:
Executive functioning inhibition | 16 weeks, + 6 months
  Stroop test
Executive functioning: task switching | 16 weeks, + 6 months
  Trail Making A-B
Executive functioning updating | 16 weeks, + 6 months
  letter memory task
Fluid intelligence | 0 weeks, for baseline
  Matrix reasoning (WAIS test)
Self-reported measure | 0 and 16 weeks, + 6 months
  Nijmegen CI Questionnaire (NCIQ): 5-points scale assesses communication and quality. of life in persons with a cochlear implant. There are 6 subdomains, ranging from 0 (low) to 100 (high). Subdomains are evaluated by adding together the scores of each questions per subdomain and dividing this by the number of completed items per subdomain. A total score is reported.
Self-reported measure | 0 weeks, for baseline
  Coping: Utrechtse Coping Lijst: A validated questionnaire based on a 4-point scale: assesses coping strategies in daily life. There are 7 subscales and 1 total score. Scale varies between 1 (low) and 4 (high).
Transfer of change in speech in noise intelligibility | Change at 6 months post intervention compared to primary outcome
  LIST sentences presented in speech-weighted noise. Participants are required to repeat sentences in noise. The Leuven Intelligibility Sentences Test (LIST, (van Wieringen & Wouters, 2008)) was specifically designed for speech perception in noise assessment in CI users. The test has a high test-retest reliability and a steep slope making it very sensitive to small improvements in performance.
  An improvement of 2dB results in a clinically relevant improvement in speech.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid van Wieringen, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Experimental ORL, Dept Neurosciences, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magits S, Boon E, De Meyere L, Dierckx A, Vermaete E, Francart T, Verhaert N, Wouters J, van Wieringen A. Comparing the Outcomes of a Personalized Versus Nonpersonalized Home-Based Auditory Training Program for Cochlear Implant Users. Ear Hear. 2023 May-Jun 01;44(3):477-493. doi: 10.1097/AUD.0000000000001295. Epub 2022 Oct 29. PMID 36534665
- [Derived] van Wieringen A, Wouters J. Lilliput: speech perception in speech-weighted noise and in quiet in young children. Int J Audiol. 2023 Aug;62(8):747-755. doi: 10.1080/14992027.2022.2086491. Epub 2022 Jun 22. PMID 35732012